CLINICAL TRIAL: NCT00328224
Title: Oral Status and Prevalence of Dental Trauma in Children Treated With Ritalin Due to Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 230606-HMO-CTIL
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2006-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Dental Caries; Dental Occlusion, Traumatic
Keywords: ritalin; ADHA; dental status; periodontal status; Attention-Deficit Hyperactivity Disorder; Dental trauma
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dental Caries; Dental Occlusion, Traumatic

STUDY DESIGN:
Observational Model: Case-Control

SUMMARY:
To evaluate the dental status of children using ritalin and suffering from ADHA in comparison to healthy children.

DETAILED DESCRIPTION:
In this trial oral and dental status of 30 children (ages 5-12) who suffer from ADHD and treated with ritalin will be evaluated. Parameters that will be checked are the following: DMFT - decay, missing, filling teeth for dental status, GI - gingival index, PI - plaque index for periodontal status. OJ - over jet and OB - over bite for inter-maxillary relations and susceptibility for dental trauma. In addition these parameters will be collected for 30 age and sex match healthy children.

ELIGIBILITY:
Inclusion Criteria:

* children ages 5-12 years healthy children children taking ritalin who suffer from ADHD

Exclusion Criteria:

* all others

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children children with adhd treated with ritalin
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-05; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ram, DMD, Principal Investigator — Hadassah Medical Organization; Meir Redlich, DMD,PhD, Study Director — Hadassah Medical Organization; Hadas Katz-Sagi, DMD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel